CLINICAL TRIAL: NCT01629251
Title: Closing the Loop for 36 Hours in Adolescents With Type 1 Diabetes: Evaluation of Reduced Meal Bolusing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Principal Research Associate, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DAN02
Record Dates: First submitted 2011-04-05; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Type 1 Diabetes
Keywords: Closed-loop insulin delivery; Post-prandial hypoglycaemia; Meal insulin dosing
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed-loop with standard meal insulin bolus (Active Comparator): Subcutaneous basal insulin delivery will be adjusted following the advice by a computer-based algorithm, based on subcutaneous sensor glucose readings. Standard meal insulin dosing will be performed at each meal, following individual standard clinical practice.
  Interventions: Device: Closed-loop insulin delivery
- Closed-loop with reduced meal insulin bolus (Experimental): Subcutaneous basal insulin delivery will be adjusted following the advice by a computer-based algorithm, based on subcutaneous sensor glucose readings. The standard meal insulin dose will be reduced by 20 to 50%.
  Interventions: Device: Closed-loop insulin delivery

INTERVENTIONS:
Device: Closed-loop insulin delivery — Subcutaneous basal insulin delivery will be adjusted following the advice by a computer-based algorithm, based on subcutaneous sensor glucose readings. Standard or reduced meal insulin dosing will be performed in a randomised design.

SUMMARY:
The main focus of our research is the development of a closed-loop system for glucose control in people with type 1 diabetes. After having demonstrated the safety and efficacy of overnight closed-loop insulin delivery, we are extending the evaluation of closed-loop to the daytime. Meal-related insulin dosing can be challenging and prandial insulin overdosing can be associated with the occurrence of postprandial hypoglycaemia, thus representing a confounding factor of hypoglycaemia free glucose control during the day. A further investigation is needed to evaluate alternative strategies for prandial insulin dosing. We will study eight adolescents with type 1 diabetes during closed-loop insulin delivery combined with either standard or reduced insulin doses with the meals, in a randomised crossover design. Stable glucose isotopes will be administered to collect data for modelling of glucose turnover around the meals, during daily activities and overnight.

The information provided by the use of glucose isotopes would be very helpful to increase our understanding of the physiology of glucose turnover and to facilitate the development of an improved control algorithm. Ultimately this study will help with the development of a closed-loop system to match insulin infusions to change in glucose levels in real life conditions.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 12 and 18 years of age (inclusive).
* The subject has had type 1 diabetes, as defined by WHO for at least 1 year or is confirmed C-peptide negative.
* The subject will have been on insulin pump user for at least 3 months, with good knowledge of insulin self-adjustment.
* HbA1c ≤ 12 % based on analysis from central laboratory

Exclusion Criteria:

* Non-type 1 diabetes mellitus including those secondary to chronic disease
* Any other physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results
* Current treatment with drugs known to interfere with glucose metabolism such as systemic corticosteroids, non-selective beta-blockers and MAO inhibitors
* Known or suspected allergy against insulin
* Subjects with clinical significant nephropathy, neuropathy or proliferative retinopathy as judged by the clinician
* Total daily insulin dose >= 2 IU/kg
* Post-menarchal girls who are pregnant or intending to become pregnant or are breastfeeding
* Any coexisting cardiac and respiratory condition

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint | 36hours
  The primary outcome measure is time spent with plasma glucose concentration in the target range (3.9-10.0mmol/L) between 24:00 on Day 1 and 08:00 on Day 3 (32 hours) as obtained with closed-loop insulin delivery in comparison with conventional insulin pump therapy.

SECONDARY OUTCOMES:
Secondary efficacy endpoints | 36 hours
  * Total and basal insulin delivery between 24:00 on Day 1 and 08:00 on Day 3 (36 hours)
  * CGM glucose levels between 24:00 on Day 1 and 08:00 on Day 3 (36 hours)
  * Overnight glucose levels between 24:00 on Day 1 and 08:00 on Day 2 (8 hours), and between 24:00 on Day 2 and 08:00 on Day 3 (8 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Wellcome Trust Clinical Research Facility, Addenbrooke's Hospital, Cambridge, United Kingdom

REFERENCES:
- [Background] Hovorka R, Allen JM, Elleri D, Chassin LJ, Harris J, Xing D, Kollman C, Hovorka T, Larsen AM, Nodale M, De Palma A, Wilinska ME, Acerini CL, Dunger DB. Manual closed-loop insulin delivery in children and adolescents with type 1 diabetes: a phase 2 randomised crossover trial. Lancet. 2010 Feb 27;375(9716):743-51. doi: 10.1016/S0140-6736(09)61998-X. Epub 2010 Feb 4. PMID 20138357